CLINICAL TRIAL: NCT00814762
Title: Study to Evaluate the Safety and Reactogenicity of the HIV Vaccine SB732462 in HIV Infected Subjects Aged 18 to 55 Years Old
Brief Title: Safety of the HIV Vaccine 732462 in HIV Infected Subjects Aged 18 to 55 Years Old
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 112353
Record Dates: First submitted 2008-12-23; First posted 2008-12-25 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: AIDS
Keywords: immunogenicity; HIV; reactogenicity; safety; vaccine; HIV Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- HIV 732462 Group (Experimental): Subjects received 2 doses of the HIV Vaccine 732462 into the deltoid muscle of the dominant arm, on a 0, 1 Month schedule.
  Interventions: Biological: HIV Vaccine 732462
- Placebo Group (Placebo Comparator): Subjects received 2 doses of the placebo vaccine into the deltoid muscle of the dominant arm, on a 0, 1 Month schedule.
  Interventions: Biological: Placebo vaccine

INTERVENTIONS:
Biological: HIV Vaccine 732462 — Two doses reconstituted adjuvanted vaccine, injected intramuscularly, at an interval of approximately one month.
  Arms: HIV 732462 Group
Biological: Placebo vaccine — Two doses of placebo, injected intramuscularly, at an interval of approximately one month
  Arms: Placebo Group

SUMMARY:
The purpose of this research study is to evaluate the safety of GSK Biologicals' investigational HIV vaccine 732462, administered as two doses approximately 1 month apart, in a small group of HIV infected people.

DETAILED DESCRIPTION:
This multicenter observer-blind study will determine the safety and reactogenicity of GSK Biologicals' investigational HIV vaccine 732462 in two sequentially enrolling cohorts of HIV-infected subjects treated with HAART (highly active antiretroviral therapy) and HIV infected treatment naïve subjects, respectively.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy the following criteria at screening and before vaccination:

* A male or female, aged between and including 18-55 years at the time of first vaccination.
* Known to be HIV-1 infected and under care of an HIV physician for a minimum of 6 months. However, subjects who initially presented with primary HIV infection need to have been diagnosed and under care for 12 months.
* Written informed consent obtained from the subject prior to any study procedure.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* If the subject is female, she must be of non-childbearing potential, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions throughout the duration of the study.
* CD4 count ≥ 450 cells per mm³

Additional inclusion criteria for subjects enrolled in the first cohort (HIV-infected subjects receiving HAART):

* Stable on highly active antiretroviral therapy (HAART) for at least one year.
* Undetectable viral load

Additional inclusion criteria for subjects enrolled in second cohort (treatment-naïve HIV-infected subjects):

* HAART-naïve (never received anti-retrovirals after HIV diagnosis)
* VL 5000-80000 copies/mL at screening
* Commencement of HAART is not expected based on current assessment within next year.

Exclusion Criteria:

The following criteria should be checked at the time of screening and before vaccination. If any apply, the subject must not be included in the study:

* Infection with HIV-2
* Had an AIDS defining illness (CDC Classification).
* Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding the first dose of study vaccine/placebo, or planned use of any investigational or non-registered product other than the study vaccine during the study period.
* Drug therapy with immunomodulators or steroids within the three months preceding the first dose of study vaccine/placebo or planned administration during the study period
* Administration of immunoglobulins and/ or any blood products within the three months preceding the first dose of study vaccine/placebo or planned administration during the study period.
* Planned administration of a vaccine not foreseen by the study protocol during the period starting 30 days before the first dose of study vaccine/placebo and ending at Month 4 It is recommended that the vaccination history of all subjects has been reviewed with their health care provider and that they have been encouraged to be fully vaccinated according to their country vaccination schedule for HIV- infected persons before enrolment into this study.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Any previous vaccination or immunotherapy against HIV.
* History of immune reconstitution disease when commencing antiretroviral therapy (for HIV-infected subjects receiving HAART)
* A family history of hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute or chronic infective hepatitis (A past history of hepatitis B or C is not an exclusion criterion).
* Acute or chronic, clinically relevant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Any condition (including alcohol and drug abuse) which, in the opinion of the investigator, could compromise the subject's safety or adherence to the study protocol
* History of medically confirmed autoimmune disease
* History of malignancy, other than squamous cell or basal cell skin cancer, unless there has been surgical excision that is considered to have achieved cure
* Asthma requiring daily steroid or long acting ß agonist prevention
* Unstable asthma defined as:

  * Sudden acute attacks occurring in less than three hours without an obvious trigger.
  * Hospitalisation for asthma in the last two years
* Food or wine induced asthma
* Known sensitivity to sulfites or aspirin
* Known sensitivity to aminoglycoside antibiotics

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2009-02-03 (Actual); Primary Completion 2010-08-18 (Actual); Study Completion 2010-08-18 (Actual)

PRIMARY OUTCOMES:
Number of subjects with solicited local symptoms | During a 7-day follow-up period after each vaccination (i.e. the day of vaccination and 6 subsequent days)
  Assessed solicited local symptoms were: pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain causing inability to perform usual social and functional activities. Grade 1 redness/swelling = redness/swelling spreading beyond (>) 50 millimeters (mm) of injection site.
Number of subjects with solicited general symptoms | During a 7-day follow-up period after each vaccination (i.e. the day of vaccination and 6 subsequent days)
  Assessed solicited general symptoms were abdominal pain, anorexia, diarrhoea, fatigue, headache, myalgia, nausea, sweating, vomiting and temperature [oral temperature equal to or above (≥) 37.7 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptoms = symptoms causing inability to perform usual social and functional activities. Grade 3 anorexia = loss of appetite associated with significant weight loss. Grade 3 diarrhoea = bloody diarrhoea or increase of ≥7 stools per 24 hour period, or IV fluid replacement. Grade 3 nausea/vomiting = persistent nausea/vomiting resulting in minimal oral intake for more (>) than 48 hours/in orthostatic hypotension or aggressive rehydration indicated. Grade 3 temperature = temperature between 39.4- 40.5 °C
Number of subjects with unsolicited Adverse Events (AEs) | Day 0-Day 29 after each vaccination
  An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Number of subjects with Serious Adverse Events (SAEs) and medically attended visits | From Screening at Day -42 and up to the additional visit post study end, Month 12
  Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Medically attended visits include any kind of medical attention such as hospitalization, an emergency room visit or a visit to or from medical personnel (medical doctor) for any reason.
Number of subjects with study pre-defined Human Immunodeficiency Virus (HIV)-related adverse events | From Day 0 to study end at Month 12
  Study pre-defined HIV-related AEs included: cluster of differentiation-4 (CD4) count decrease [(≥)25% post vaccination], viral load increase [(≥)50 copies per (/) milliliter (mL) of HIV ribonucleic acid (RNA) post-vaccination, for cohort A and at least 0.5 log post-vaccination for cohort B], initiation of Highly Active Anti-Retroviral Therapy (HAART) for cohort B, or changes in HAART for cohort A, abnormal biochemistry and haematology parameters.
Number of subjects presenting abnormal biochemical and haematological values (any and grade ≥ 3) | From Day 0 to study end at Month 12
  Assessed biochemical and haematological parameters included: Absolute neutrophil count (ANC), Haemoglobin (Hgb), Partial Thromboplastin Time (PTT), Platelets decreased (PLT/D), WBC decreased (WBC/D), Albumin serum low (ALB/SL), Alkaline Phosphatase (ALP), Alanine aminotransferase (SGPT), Aspartate aminotransferase (SGOT), Bilirubin Total (BL/T), Creatinine (CRT), Potassium serum high (K/SH), Potassium serum low (K/SL), Sodium serum high (Na/SH), Sodium serum low (NA/SL), Uric acid (UA).
Time to initiation of HAART therapy (for treatment-naïve HIV-infected subjects) or change in HAART therapy (for HIV-infected subjects receiving HAART) | From Day 0 to Month 12
  Time to HAART initiation and/or HAART changes was expressed in days from administration of first dose.

SECONDARY OUTCOMES:
CD4 count and change of CD4 count from baseline | From Day 0 to Month 12
  Baseline was defined as the value measured in the pre-vaccination blood sample obtained at Day 0 prior to the administration of the first dose.
Viral load and change in viral load from baseline | From Day 0 to Month 12
  Baseline was defined as the value measured in the pre-vaccination blood sample obtained at Day 0 prior to the administration of the first dose.
Cluster of differentiation 40 ligand (CD40L+) CD4+ T-cell-mediated immune response (as measured by ICS) | Months 0, 4, 12 and at Day 44
  CD40L+ and CD4+ T cell immune response was assessed via Intracellular Cytokine Staining (ICS) and included: breadth which was by looking at response to at least 1, 2, 3 antigens and to all 4 antigens [p17, p24, Necrosis Factor (Nef) and Reverse Transcriptase (RT)], intensity which was defined as frequency of the 4 antigent-specific CD40L+CD4+ T cells expressing at least Interleukin 2 (IL-2) or Tumor Necrosis Factor alpha (TNFa) and/or Interferon gamma (INFg) and cytokine co-expression profile defined as the frequency of the 4 antigen-specific CD40L+CD4+ Tcells expressing IL-2 and/or TNFa and/or IFNg.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Germany (5):
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg

REFERENCES:
- [Derived] Harrer T, Plettenberg A, Arasteh K, Van Lunzen J, Fatkenheuer G, Jaeger H, Janssens M, Burny W, Collard A, Roman F, Loeliger A, Koutsoukos M, Bourguignon P, Lavreys L, Voss G. Safety and immunogenicity of an adjuvanted protein therapeutic HIV-1 vaccine in subjects with HIV-1 infection: a randomised placebo-controlled study. Vaccine. 2014 May 7;32(22):2657-65. doi: 10.1016/j.vaccine.2013.10.030. Epub 2013 Oct 19. PMID 24144472
- See also: Results for study 112353 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/112353?search=study&b%22b''%22#rs